CLINICAL TRIAL: NCT00822055
Title: Comparison of the Fixed Combinations of Brimonidine/Timolol and Dorzolamide/Timolol in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COM0501
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Brimonidine Tartrate; Timolol; Brimonidine Tartrate, Timolol Maleate Drug Combination; dorzolamide; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): brimonidine/timolol Fixed-combination monotherapy
  Interventions: Drug: brimonidine tartrate 0.2%/timolol maleate 0.5% fixed combination
- 2 (Active Comparator): dorzolamide/timolol fixed-combination monotherapy
  Interventions: Drug: dorzolamide hcl 2%/timolol maleate 0.5% fixed combination
- 3 (Active Comparator): prostaglandin analogue + brimonidine/timolol fixed combination
  Interventions: Drug: brimonidine tartrate 0.2%/timolol maleate 0.5% fixed combination as adjunctive to current prostaglandin therapy
- 4 (Active Comparator): prostaglandin analogue + dorzolamide/timolol fixed combination
  Interventions: Drug: dorzolamide hcl 2%/timolol maleate 0.5% fixed combination as adjunctive to current prostaglandin therapy

INTERVENTIONS:
Drug: brimonidine tartrate 0.2%/timolol maleate 0.5% fixed combination — 1 drop BID in each eye
  Other Names: Combigan®
  Arms: 1
Drug: dorzolamide hcl 2%/timolol maleate 0.5% fixed combination — 1 drop BID in each eye
  Other Names: Cosopt®
  Arms: 2
Drug: brimonidine tartrate 0.2%/timolol maleate 0.5% fixed combination as adjunctive to current prostaglandin therapy — 1 drop BID in each eye
  Other Names: Combigan®
  Arms: 3
Drug: dorzolamide hcl 2%/timolol maleate 0.5% fixed combination as adjunctive to current prostaglandin therapy — 1 drop BID in each eye
  Other Names: Cosopt®
  Arms: 4

SUMMARY:
This study compares the efficacy and tolerability/comfort of brimonidine/timolol and dorzolamide/timolol in patients with open-angle glaucoma or ocular hypertension. In an investigator masked randomisation process, each subject is allocated to received either brimonidine/timolol or dorzolamide/timolol as fixed-combination monotherapy or as an adjunctive to a prostaglandin analogue for a period of 12 weeks. After screening, patient returns at baseline, Month 1 and Month 3 for ophthalmic evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years
* Female subjects of childbearing potential must have negative pregnancy test and practice contraception
* Subjects must have confirmed diagnosis of primary open-angle glaucoma or ocular hypertension in both eyes
* Subjects who are or have been insufficiently responsive to IOP reducing monotherapy and use of either study medication is deemed appropriate
* Subjects able to complete questionnaires and provide informed consent

Exclusion Criteria:

* Female subjects who are pregnant, planning to become pregnant during study period, breast feeding or not practicing a reliable method of birth control
* Subjects wherein the study drugs are contraindicated
* Subjects who have had intraocular surgery with 6 months (3 months for laser)
* Subjects with known side effects/allergy or sensitivity to any component of study treatments
* Subjects with any uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean IOP | 12 weeks

SECONDARY OUTCOMES:
Patient tolerability/comfort measured by Likert scale | Month 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Barrie, Ontario, Canada

REFERENCES:
- [Derived] Nixon DR, Yan DB, Chartrand JP, Piemontesi RL, Simonyi S, Hollander DA. Three-month, randomized, parallel-group comparison of brimonidine-timolol versus dorzolamide-timolol fixed-combination therapy. Curr Med Res Opin. 2009 Jul;25(7):1645-53. doi: 10.1185/03007990902994041. PMID 19476406